CLINICAL TRIAL: NCT07192146
Title: Patient Reported Outcomes and Associated Factors Following Endodontic Emergency Treatment: A Prospective Cohort Study
Brief Title: Patient Reported Outcomes and Associated Factors Following Endodontic Emergency Treatment
Status: Recruiting | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Other Study IDs: HREC-DCU 2023-122
Record Dates: First submitted 2025-07-20; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-07

CONDITIONS: Moderate to Severe Endodontic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to analyze the improvement of postoperative pain and Oral Health-Related Quality of Life (OHRQoL) following endodontic emergency treatment, as well as the contributing factors affecting the change including age, gender, tooth type, dental arch, pulpal status, percussion pain, radiographic evidence of periapical lesions, type of emergency treatment (pulpotomy / partial pulpectomy / complete pulpectomy), and occlusal adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Presence of moderate to severe pain as measured by a Numerical Rating Scale (NRS) score ≥ 4
* Pain of endodontic origin confirmed through clinical and/or radiographic examination

Exclusion Criteria:

* Refused or were unable to provide informed consent or complete the questionnaire
* Were currently or recently taking immunosuppressive agents, long-term anti-inflammatory medications, or antibiotics
* Had non-endodontic or mixed-origin pain
* Had already initiated endodontic treatment on the affected tooth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergo endodontic emergency treatment.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | From enrollment to the end of treatment at 2 years
  Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Oral health-related quality of life | From enrollment to the end of treatment at 2 years
  Higher scores mean a worse outcome.

OTHER OUTCOMES:
Prognostic factors associated with the improvement of postoperative pain | From enrollment to the end of treatment at 2 years
Prognostic factors associated with the improvement of oral health-related quality of life | From enrollment to the end of treatment at 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided